CLINICAL TRIAL: NCT01716026
Title: Establishment of the Initial Protocol With Intravitreal Bevacizumab for the Treatment of Choroidal Neovascularization Associated With High Myopia:3 vs 1.
Brief Title: Initial Treatment With Bevacizumab in Choroidal Neovascularization Associated to High Myopia
Acronym: BENEMCOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOBA-04-2012
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2021-06

CONDITIONS: Choroidal Subfoveal/Juxtafoveal Neovascularization in High Myopia
Keywords: high myopia; choroidal neovascularization
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 Month Load with 9 month p.r.n. (Active Comparator): 3 Monthly bevacizumab injections with 9 p.r.n. monthly doses if patient meets the treatment criteria for each monthly visit
  Interventions: Drug: Bevazizumab intravitreal injection
- Single Dose Load Phase (Experimental): Single dose treatment with bevacizumab, followed by 2 sham injections if conditions are met in the months 2 and 3, and followed with bevacizumab monthly p.r.n. as per protocol
  Interventions: Drug: Bevazizumab intravitreal injection

INTERVENTIONS:
Drug: Bevazizumab intravitreal injection — Intravitreal injection of bevacizumab
  Other Names: Avastin Injection

SUMMARY:
The purpose of this protocol is to determine wether the initial protocol in the treatment of subfoveal choroidal neovascularization associated to High Myopia with bevacizumab intravitreal injections is more effective when using 3 doses vs using 1 single dose in the load period

ELIGIBILITY:
Inclusion Criteria:

* Active subfoveal/juxtafoveal choroidal neovascularization in high myopia confirmed by Fundus Fluorescein angiography and Optical Coherence Tomography
* Best corrected visual acuity loss with less than 6 months of evolution, caused mainly by the neovascular lesion (based in investigator´s criteria)
* No atrophy or fibrotic component that may prevent visual acuity improvement
* Patients previously treated with Photodynamic Therapy are allowed to participate in this study
* Signed informed consent
* Signed data protection consent
* Negative pregnancy test in potential childbearing women at screening, with accepted contraceptive method during the whole study

Exclusion Criteria:

* Previous vitreous surgery in study eye
* Tractional maculopathy or epiretinal membrane found in Optical Coherence Tomography
* Media opacities that may prevent correct fundus assessment
* Lack of posterior capsule integrity in pseudophakic patients
* Patients with great possibilities of not being able to attend to study visits / follow visit procedures (investigator´s criteria)
* Patients previously treated with intravitreal antiangiogenic injections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) Best corrected visual acuity | 1 Year
  Differences in best corrected visual acuity in the exit visit compared to the one obtained at screening visit
Retinal thickness | 1 Year
  Retinal thickness assessed by Spectral Domain Optical Coherence Tomography
Number of total injections during study | 1 Year
  Total count of bevacizumab intravitreal injections during the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Jose Maria Ruiz-Moreno, MD PhD, Principal Investigator — University of Castilla-La Mancha
Locations (11):
- Spain (11):
  - CHUS - Fundacion IDICHUS, Santiago de Compostela, La Coruña
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Reina Sofia, Murcia
  - Hospital Virgen de Valme, Seville
  - Hospital Virgen de la Macarena, Seville
  - Hospital General Universitario de Valencia, Valencia
  - IOBA - Instituto Universitario de Oftalmobiologia Aplicada, Valladolid
  - Hospital Universitario Rio Hortega, Valladolid